CLINICAL TRIAL: NCT03497416
Title: Preoperative Anemia Among the Elderly Undergoing Major Abdominal Surgery: Impact on Healthcare Outcomes
Brief Title: Impact of Preoperative Anemia on Healthcare Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: PANAMA
Record Dates: First submitted 2018-03-25; First posted 2018-04-13 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Anemia
Keywords: Preoperative Anemia; elderly; healthcare outcomes
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anemic
  Interventions: Other: No intervention
- Non-anemic
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Preoperative anemia is a known risk factor for morbidity, mortality and increased healthcare resource utilisation. The Investigator's previous study demonstrated the rate of preoperative anemia in Singapore General Hospital (SGH) to be at 26.6%. The rate is highest in the elderly group which stands at 49.9%. The main objective of this study is to investigate the perioperative morbidity and mortality, blood transfusion rate, healthcare outcomes and patient-centric outcomes among anemic elderly patients undergoing major surgery. The investigators hypothesize that elderly patients who undergoes major abdominal surgery with preoperative anemia will have higher composite morbidity and mortality rates (primary outcome), longer length of hospital stay, higher blood transfusion requirements and lower health-related quality of life (HRQoL) at 1, 3 and 6 months (secondary outcomes) when compared to elderly patients without preoperative anemia. The investigators will conduct a prospective observational study of 450 consecutive patients above 65 years, who are undergoing elective major open abdominal surgery in SGH over 12 months. Baseline clinical assessment, including iron studies for anemic patients, will be done within 14 days prior to surgery. To determine the primary outcome, patients will be followed up prospectively for 30 days from the day of surgery. This will be done via a mixture of medical records review and phone interview. For secondary outcomes, the length of hospital stay and readmissions for any reason within 3 and 6 months will be recorded.

HRQoL questionnaires will be done through phone calls by a study team member. Findings from this study will hopefully fill the knowledge gaps such as how anemia impacts elderly people in terms of perioperative morbidity, mortality, postsurgical quality of life and their eventual return to the community as well as providing local data on the healthcare resource utilisation in this group.

DETAILED DESCRIPTION:
Preoperative anemia is a common and important problem in the elderly.

Many studies have established association between preoperative anemia and poor postoperative outcomes. Some propose that preoperative anemia is an independent risk factor of adverse outcomes. Preoperative anemia is also one of the strongest predictors of perioperative blood transfusion which is independently associated with increased risk of perioperative morbidity and mortality. Consequently, preoperative anemia increases healthcare utilization and costs due to increased blood transfusion requirements, prolonged length of hospital stay and hospital readmission rates. As more elderly patients undergo surgery yearly, there is a need to improve perioperative outcome, contain healthcare costs and help rapid return to community. Addressing preoperative anemia could be one such strategy as it may lead to decreased need for blood transfusion, and reduction of morbidity and mortality, and improved health-related quality of life. The relationship between anemia and quality of life is well documented in patients with cancer and with end-stage renal failure, but not so well examined in elderly postoperative patients.

The primary aim of this study is to investigate the impact of preoperative anemia on postoperative complications as defined by presence of Postoperative Morbidity Survey (POMS) defined complications at day 5. The 9 domains within POMS allow classification of complications into various organ categories, such as cardiac, respiratory, infectious etc. The secondary aim of this study is to investigate the impact of preoperative anemia on the severity of post operative complications as classified with the Clavien Dindo Classification and Comprehensive Complication Index.

Other secondary aims of this study include investigating the association between preoperative anemia and length of hospital stay, readmission within 6 months, days alive and out of hospital (DaOH) within 6 months, and 30-day mortality. Data generated on the potential healthcare costs of this modifiable risk factor would help to provide the background for future studies on intervention strategies and its cost effectiveness.

Another secondary aim of the study is to examine the relationship between preoperative anemia and baseline and postoperative health-related quality of life indices up to 6 months postoperative using the EQ-5D questionnaire. The results of this study will encourage policies that risk profile patients who may require extra support on returning to the community. In the longer term, the investigators hope to spur studies which look at the optimal hemoglobin level prior to hospital discharge after surgery.

Significance of the Study

The findings from this study will have a significant impact on the way clinicians and researchers approach preoperative anemia in the elderly. The full clinical, patient-centred, and economic impact of operating on an anemic elderly patient has not been clearly elucidated, especially in the local context. In the longer term, this study may set the foundation for nationwide policies to address anemia in the surgical population with the aim of improving patient outcomes in the most cost effective manner.

ELIGIBILITY:
Inclusion Criteria:

1. At least 65 years of age and signed written informed consent.
2. Patients undergoing elective major open abdominal surgery for benign or malignant disease.

Exclusion Criteria:

1. Transplantations (specifically patients who are admitted to the hospital for a transplantation and has a transplantation procedure and any additional surgical procedure during the hospitalisation will be excluded; any operation done after the patient has been discharged from the transplantation stay will be included)
2. Inability to comprehend and/or perform study procedures in the investigator's opinion.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly at least 65 years of age who are undergoing elective major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Preoperative anemia and morbidity | 5 days from surgery
  To determine the association between preoperative anemia and morbidity at the 5th postoperative day (POD) as indicated by presence of any Post-Operative Morbidity Survey (POMS) defined complications.

SECONDARY OUTCOMES:
Preoperative anemia and 30-day morbidity using POMS | 1 month from index surgery
  To determine the association between preoperative anemia and trend of POMS-defined complications for the first 30 post-operative days
Preoperative anemia and 30-day morbidity using Comprehensive Complication Index | 1 month from index surgery
  To determine the association between preoperative anemia and severity of postoperative complications within 30-days postoperatively using the Clavien Dindo Classification system (CDC) and Comprehensive Complication Index (CCI).
Preoperative anemia and mortality | 1 month from index surgery
  To determine the association between preoperative anemia and incidence of 30-day mortality

OTHER OUTCOMES:
Preoperative anemia and patient's health related quality of life (HRQoL) | 1,3 and 6 months from index surgery
  To determine the association between preoperative anemia and HRQoL as demonstrated by the EQ-5D scores at baseline, 1, 3 and 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hairil R Abdullah, MMed, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No